CLINICAL TRIAL: NCT06888596
Title: Feasibility of High-intensity Interval Training in Older Adults with HIV and Co-Occurring Hypertension
Brief Title: Feasibility of HIIT in Older Adults with HIV and Hypertension
Acronym: HARC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Raymond Jones, Assistant Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB-300009214; UWSC14238 (Other Grant/Funding Number: University of Washington)
Record Dates: First submitted 2025-03-13; First posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: HIV; Hypertension; Exercise
Keywords: HIIT
MeSH Terms: conditions — Hypertension; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- High-Intensity Interval Training (Experimental): Participants will follow a HIIT program adapted from previously successful exercise interventions. Participants will attend 2-weekly sessions of HIIT training for 6 weeks for a total of 12 visits. We have previously established commitments in other high-risk clinical populations, and are confident that we can ensure a moderate adherence rate in the current study population. Intensity is based on age-predicted HR max. Each session was performed using cycle ergometer. 4 sets of 4-minute HIIT at 80-90% HR max with 3 sets of 3-minute active recovery intervals at 60-70% HR max. This is followed by a final 5-minute cool-down.
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — Exercise using cycle ergometer
  Other Names: HIIT

SUMMARY:
The goal of this HIV and Aging Pilot Program Proposal is to foster interdisciplinary collaborations in HIV and geroscience by providing emerging researchers with experience and mentorship in translational research. The focus is on collecting data on the efficacy and feasibility of short-term high-intensity interval training among older people with HIV (PWH) and co-occurring hypertension.

Non-AIDS defining comorbidities are increasingly prevalent among aging PWH. The use of antiretroviral therapies (ART) has extended life expectancy, presenting unique risks for aging-related multimorbidities. Hypertension, affecting over 50% of HIV-infected adults in the U.S., is a significant chronic disorder among PWH. Regular exercise improves function and prevents decline in adults with comorbidities. Functional outcomes are good predictors of cardiovascular health in older PWH with hypertension. Exercise improves cardiovascular, metabolic, and functional measures in young PWH, but older PWH often do not meet physical activity guidelines due to barriers like motivation, time, and pain.

The impact of high-intensity exercise on physical function in older PWH is unknown, despite evidence of benefits from low-moderate intensity exercise. Assessing the feasibility and acceptability of high-intensity exercise in older PWH with hypertension will provide valuable information for future studies.

The specific aims of the proposed study are to assess the integrity of the study protocol, including safety, adherence, and retention, to develop standard operating procedures for future trials, while determining participant perceived benefits and barriers. Additionally, the study aims to assess the variance of secondary outcomes and the effects of the intervention on the 6-minute walk test, lower extremity function as assessed by the Short Physical Performance Battery, skeletal muscle strength and endurance as assessed by isokinetic muscle testing, chronic pain evaluated by the Brief Pain Inventory and Pain assessments, markers of vascular health such as arterial stiffness, and circulating indices of inflammation including inflammatory profile, skeletal muscle degradation, and metabolism.

DETAILED DESCRIPTION:
Life expectancy for people with HIV (PWH) has increased in the antiretroviral therapy (ART) era and shifted the demography of the HIV epidemic toward the aging population. By the year 2030, an estimated 70% of PWH in the United States will be at least 50 years of age, thus implicating age-related comorbidities as a potential challenge for PWH. In particular, hypertension represents a major co-morbidity burden among PWH. Regular physical activity improves function in adult populations with comorbidities and prevents functional declines.

Maintenance of functional status, determined by measures of physical performance, is a good predictor of cardiovascular outcomes among older PWH with co-occurring hypertension. Exercise is the only intervention with evidence to support its use in treating age-related functional declines. Exercise is a strategy employed by PWH and rehabilitation professionals to address the functional decline and improve the health and quality of life of those individuals. Exercise interventions in PWH support the evidence that exercise can improve cardiovascular, metabolic, and functional measures in younger PWH. Though meeting the recommended guidelines for regular physical activity in older adults is feasible, the repercussions of high-intensity interval training in improving physical function are unknown despite evidence displaying functional improvements following low and moderate-intensity interventions.

While many exercise studies have reflected the benefit of six to twelve weeks of exercise, many report that the results are limited to the participants who are motivated with good compliance and completion profiles. In real-world situations, adherence to exercise, particularly high-intensity exercise, may fall below desirable levels and hinder the effectiveness of the programs. This may be due, in part, to perceived benefits and barriers to exercise in older PWH. Despite the growing body of research aimed at determinants of adherence to pharmaceutical treatment, adherence to exercise among PWH remains an under-researched area.

The purpose here is to evaluate the efficacy and efficacy of a high-intensity interval training intervention for improving the physical function of older PWH and co-occurring hypertension. The central hypothesis is that high-intensity exercise will improve functional decrements of older PWH. An evaluation of high-intensity interval training in PWH may be important as this population has impairment in functional outcomes compared with age-matched uninfected controls, with even greater impairments among older PWH. Underlying inflammation, pain, and skeletal muscle degradation related to HIV suggest that older PWH may require higher doses of exercise to restore or achieve levels of physical function. Thus, the objective of this pilot application is to evaluate the efficacy and feasibility of short-term high-intensity interval training among 15-20 older PWH > 50 years with co-occurring hypertension, recruited from CNICS. To achieve this objective, the investigators propose to conduct a pilot study to address the following specific aims, which are crucial to designing future studies:

Specific Aim 1: To assess the integrity of the study protocol, including safety, adherence to the interventions, and retention to study visits, in order to develop standard operating procedures for guidance of a future trial. Additionally the investigators will determine participant perceived benefits and barriers, assessed by the Exercise Benefits and Barriers Scale.

Specific Aim 2: To assess the variance of secondary outcomes and effects of the intervention on outcomes including 1) 6-minute walk test, 2) lower extremity function, assessed by the Short Physical Performance Battery (SPPB), 3) skeletal muscle strength and endurance, assessed by isokinetic muscle testing, 4) chronic pain, evaluated by the Brief Pain Inventory and Pain assessments, 5) markers of vascular health (e.g., arterial stiffness), 6) circulating indices of inflammation (e.g. inflammatory profile [IL-1β, TNF-α, IL-6, CRP, IL-8, IL-10], skeletal muscle degradation [creatine kinase], and metabolism [fasting glucose, HA1C, lactate, and fasting cholesterol].

ELIGIBILITY:
Inclusion Criteria:

* >= 50 years of age at study entry
* must be on ART regimen
* Inactive Lifestyle (<150 minutes per week of moderate activity on CHAMPS Questionnaire)
* CD4 T-cell count greater than 200 cell/mm^3 (
* Hypertensive (untreated SBP >=130mmHg or DBP >=80 mmHg)
* Functional limitations inhibiting the ability to exercise.

Exclusion Criteria:

* BP >140/90 despite the use of 4+ antihypertensive medications
* chronic kidney disease
* severe cardiac condition (CHF, stenosis, history of cardiac arrest, defibrillator, angina)
* Ischemic heart disease
* self reported >= 90 days of daily opioid use
* Beta Blocker Significant cognitive impairment

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2022-06-02 (Actual); Primary Completion 2024-02-21 (Actual); Study Completion 2024-02-21 (Actual)

PRIMARY OUTCOMES:
Feasibility and Acceptability | From enrollment to the end of treatment at 6 weeks
  Feasibility and acceptability was assessed by collecting data on recruitment and retention rates, intervention adherence rates, number of eligible participants required to recruit to sample size, rate of completion of the intervention (i.e., number of participants who complete all aspects of the intervention), and completion rates.

SECONDARY OUTCOMES:
Blood Pressure | From enrollment to the end of treatment at 6 weeks
  Blood pressure was assessed using oscillometry following quiet rest.
Perceived Benefits and Barriers to Exercise | Baseline and 6 weeks
  The Exercise Barriers and Benefits Scale was developed to assess people's perceptions on exercise and benefits barriers to exercise. The instrument has a four-response, forced-choice Likert-type format with responses ranging from 1 ('Strongly Disagree') to 4 ('Strongly Agree'). Scores on the total instrument can range from 43 to 172, where the higher the score, the more positively the individual perceives exercise. Additionally, the EBBS is separated into a 29-item Benefits Scale and a 14-item Barriers scale.
Rating of Perceived Exertion | Week 1-6 of Intervention
  measured using the Borg RPE 6-20 Scale
Body Mass Index | From enrollment to the end of treatment at 6 weeks
  Body mass index was assessed using height and weight at baseline and post-intervention.
Cardiorespiratory Fitness | From enrollment to the end of treatment at 6 weeks
  Cardiorespiratory fitness was assessed using the fast-paced 6-minute walk test
Physical Function | From enrollment to the end of treatment at 6 weeks
  SPPB was performed as a measure of functional status through the domains of balance, strength, and gait measurements. The balance tests consisted of standing static balance in three positions; lower limb strength through sit-to-stand from a chair; and walking speed at a normal pace (4-meter walk test). Each test is scored from 0 (inability to perform the task) to 4 points (best performance) with total SPPB scores ranging from 0 to 12 points across all tasks.

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Jones, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No
These data are very preliminary and thus exploratory in nature. This was used to build a larger intervention. However, should researchers request information, we will disseminate IPD as deemed necessary.